CLINICAL TRIAL: NCT03653858
Title: Controlled Randomized Clinical Trial to Assess Efficacy of Deep Brain Stimulation (DBS) of the slMFB in Patients With Treatment Resistant Major Depression
Brief Title: Efficacy Study of Deep Brain Stimulation in Patients With Treatment Resistant Major Depression
Acronym: FORESEE III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, Prof. Dr., Principal Investigator, Head of Interventional Biological Psychiatry, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P000767; DRKS00014947 (Registry Identifier: German Clinical Trials Register); CIV-17-07-020746 (Other: Eudamed Number)
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Treatment-resistant Depression
Keywords: Deep Brain Stimulation; Treatment-resistant depression; Medial forebrain bundle
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, sham-controlled, double blind (patient and observer blinded)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: DBS onset in week 1 (Experimental): Implantation of Vercise GEVIA deep brain stimulation (DBS) system. DBS onset in week 1.
  2ND STAGE: After 6 months DBS ON, patients will be assessed whether they are responders or non-responders. In the subgroup of eligible responders, patients will be randomized to either DBS OFF* (for max. 3 months) or continued DBS for another 6 months. *DBS OFF until worsening of clinical depression, event (defined as > 5 points augmentation in MADRS in two consecutive visits) or for a maximum of 3 months. After DBS OFF, re-onset of DBS will be performed, followed by 6 months continuous DBS.
  Non-responders will also receive another 6 months DBS therapy in the 2nd stage. At sites other than Freiburg/Bonn, the 2nd stage consists of 6 months DBS therapy only.
  Interventions: Device: Vercise GEVIA deep brain stimulation (DBS) system
- Group B: DBS off, followed by DBS onset in week 17 (Sham Comparator): Implantation of Vercise GEVIA deep brain stimulation (DBS) system. 4 months OFF after implantation followed by DBS onset in first week of month 5.
  2ND STAGE: See group A.
  Interventions: Device: Vercise GEVIA deep brain stimulation (DBS) system

INTERVENTIONS:
Device: Vercise GEVIA deep brain stimulation (DBS) system — DBS to the superolateral branch of the Medial Forebrain Bundle (slMFB)

SUMMARY:
The primary objective of this multicenter, randomized, sham-controlled, double blind (patient and observer blinded) clinical trial is to assess the antidepressant effect of Deep Brain Stimulation (DBS) in patients with treatment resistant major depression using the Boston Scientific implantable Vercise™ GEVIA™ DBS system compared to sham.

DETAILED DESCRIPTION:
The main objective of this clinical trial is to assess the putative antidepressant efficacy of a therapeutic method called Deep Brain Stimulation (DBS) in patients suffering from severe, treatment-resistant depression, i.e. in patients who have not sufficiently improved under established antidepressant therapies (such as psychotherapy, antidepressant drug therapy, and electroconvulsive therapy).

DBS, also known as "brain pacemaker" therapy, is a neurosurgical therapeutic method that is widely established for the treatment of other conditions such as Parkinson's disease. However, DBS is not yet approved for the treatment of patients with depression.

In order to initiate DBS treatment, a neurosurgical procedure is performed in which electrodes are placed in a brain region termed 'medial forebrain bundle' (MFB). The electrodes are then used to stimulate this region with electric pulses. From previous investigations and studies with small numbers of patients, it is believed that DBS might have a positive effect on depressive symptoms in patients treated with the method.

ELIGIBILITY:
Inclusion Criteria:

1. Major depression (MD), severe, unipolar, or bipolar in an acute depression episode.
2. German mother tongue or fluent.
3. Male or female patients ≥20 and ≤75 years.
4. Hamilton Depression Rating Scale (HDRS-28) score of >21.
5. Global Assessment of Function (GAF) score of <45.
6. At least 4 episodes of depression or one chronic episode >2 years.
7. Failure to respond to

   1. adequate trials of primary antidepressants from at least 3 different classes (>5 weeks at the maximum recommended or tolerated dose) and
   2. adequate trials of augmentation/combination of a primary antidepressant (>3 weeks at the usually recommended or maximum tolerated dose) using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) and
   3. an adequate trial of electroconvulsive therapy (ECT) (>6 treatments) and an adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
8. Able to give written informed consent.
9. Compliance to participate in the study.
10. Drug free or on stable drug regimen at least 6 weeks before study entry.

Exclusion Criteria:

1. Current or past non-affective psychotic disorder.
2. Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome.
3. Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI), any contraindications to perform a planned MRI to visualize the slMFB.
4. Any surgical contraindications to undergoing DBS like deformed or displaced or not discernable target region, scarring after brain disease (infarction), need for continuous anticoagulation that cannot be bridged in order to obtain normal coagulation, present risks for anesthesia or any brain or scalp injury (even after intracranial surgery).
5. Current or unstably remitted substance abuse (aside from nicotine).
6. Pregnancy, women of childbearing age not using effective contraception and breast feeding women.
7. History of severe personality disorder.
8. Acute suicidal ideation.
9. Patients with advanced stage cardiovascular disease.
10. Patients under immunosuppressive or chemo therapy because of malignant disease.
11. Patients who had previous intracranial surgery.
12. Patients who are currently under DBS therapy or have implanted any kind of stimulator already.
13. Patients with aneurysm clips.
14. Patients with cochlear implants.
15. Patients with planned diathermy.
16. Persons who are in a relationship of dependence/employment with the sponsor or the investigator.
17. Simultaneous participation or previous participation within 30 days prior to start of screening in a clinical trial involving investigational medicinal product(s) or investigational medical device(s).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) total score | 16 weeks after surgery
  Primary outcome (Efficacy). MADRS is an established instrument to rate symptoms of depression. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts Each of the 10 items yields a score of 0 to 6. These item scores are summed up to yield a total score. The range of the total score is thus 0 to 60; higher total scores indicate more severe depressive symptoms.
  Usual cutoff points are:
  0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; >34 - severe depression
Time to Montgomery-Asberg Depression Rating Scale (MADRS) augmentation of >5 points or clinical worsening in two consecutive visits after DBS termination | Up to 3 months
  Primary outcome in 2nd stage; Description MADRS: see above.
Assessment of (Serious) Adverse Events related to Investigational Medical Device and / or surgical procedures | From IMD implantation until the end of study; assessed up to 77 weeks
  Primary outcome (Safety); (Serious) adverse events seen will be reported using standard descriptive statistical methods.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS-28) total score | 16 weeks after surgery
  HDRS is an established instrument to rate symptoms of depression. Different versions exist, using between 17 and 29 items. In this study, the 28-item version (HDRS-28) is used. The patient is rated by a clinician, items are scored either on a 3-point or 5-point Likert-type scale.
  Single item scores are summed up to yield a total score. The total score ranges from 0 to 85; a higher total score indicates more severe depressive symptoms.
Clinical Global Impression Score (CGI) total score | 16 weeks after surgery
  The CGI is a scale that measures the global severity of illness, the global improvement relative to the beginning of the study as well as the therapeutic effect and adverse reactions, score ranges from 0 to 7 for severity of illness and global improvement, a higher score indicates more severe symptoms and a worsening of symptoms; score ranges from 0 to 8 for the efficacy index, 0 means that the efficacy can't be evaluated, a score of 2 means best efficacy while a score of 8 means no therapeutic effect and more adverse reactions
Global Assessment of Functioning (GAF) total score | 16 weeks after surgery
  Score ranges from 100 (high functioning) to 1 (severly impaired)
Beck Depression Inventory (BDI-II) total score | 16 weeks after surgery
  Score ranges from 0 to 63; a higher total score indicates more severe depressive symptoms
36-Item Short Form Health Survey (SF-36) total score | 16 weeks after surgery
  Health-related quality of life questionnaire; 8 subscales: General health perceptions, physical functioning, role limitations due to physical problems, bodily pain, vitality, general mental health, role limitations due to emotional problems, social functioning. The score in each subscale ranges from 0 to 100; subscores add up to two total scores, "physical health" and "mental health", each with a score range of 0-400. Higher scores indicate better health-related quality of life.
Change over time in HDRS total score after DBS surgery with DB stimulation OFF compared to stimulation ON | assessed weekly for 16 weeks after surgery
  HDRS: see above
Change over time in CGI total score after DBS surgery with DB stimulation OFF compared to stimulation ON | assessed weekly for 16 weeks after surgery
  CGI: see above
Change over time in GAF total score after DBS surgery with DB stimulation OFF compared to stimulation ON | assessed weekly for 16 weeks after surgery
  GAF: see above
Change over time in BDI-II total score after DBS surgery with DB stimulation OFF compared to stimulation ON | assessed weekly for 16 weeks after surgery
  BDI-II: see above
Change over time in SF-36 total score after DBS surgery with DB stimulation OFF compared to stimulation ON | assessed weekly for 16 weeks after surgery
  SF-36: see above
Neuropsychological Assessments: Rey Complex Figure Test (CFT) | at 4 months after implantation
  Score range 0-36, higher scores indicate better cognitive performance
Neuropsychological Assessments: d2 concentration test (d2) | at 4 months after implantation
  Higher scores indicate better cognitive performance (total of right answers minus errors)
Neuropsychological Assessments: 5-Point-Test | at 4 months after implantation
  Score range 0-35, higher scores indicate better cognitive performance
Neuropsychological Assessments: Wechsler Adult Intelligence Scale (WAIS) (vocabulary, similarities) | at 4 months after implantation
  Score range "vocabulary": 0-32, Score range "finding similarities": 0-32, higher scores indicate better cognitive performance
Neuropsychological Assessments: Mini-Mental-Status-Test (MMST) | at 4 months after implantation
  Score range 0-30, higher scores indicate better cognitive performance
Neuropsychological Assessments: Multiple-Choice Vocabulary Intelligence Test (MWT-B) | at 4 months after implantation
  Score range 0-37, higher scores indicate better cognitive performance
Neuropsychological Assessments: Rey Visual Design Learning Test (RVDLT) | at 4 months after implantation
  Score range 0-75, higher scores indicate better cognitive performance
Neuropsychological Assessments: Word Fluency Test | at 4 months after implantation
  No maximum scores, patient has two minutes to produce answers, higher scores indicate better cognitive performance
Neuropsychological Assessments: Stroop-Test | at 4 months after implantation
  Time in s, low scores (less seconds) indicate better cognitive performance
Neuropsychological Assessments: Test for Attentional Performance (TAP) | at 4 months after implantation
  Reaction times as well as correct or false responses and omissions are measured, higher cognitive performance is indicated by fast responses, few errors and high no. of correct responses
Neuropsychological Assessments: Trail-Making Test (TMT) | at 4 months after implantation
  Time in s, low scores (less seconds) indicate better cognitive performance
Neuropsychological Assessments: Verbal Memory and Learning Ability Test | at 4 months after implantation
  Score range 0-75, higher scores indicate better cognitive performance
Neuropsychological Assessments: Hopper Visual Organization Test (VOT) | at 4 months after implantation
  Score range 0-30, higher scores indicate better cognitive performance
Neuropsychological Assessments: Digit-Span and Block-Span Test | at 4 months after implantation
  Score range 0-12 for each of for dimensions: Digit span forward, digit span backward, block span forward, block span backward. Higher scores indicate better cognitive performance
MADRS total score during long-term follow-up compared to baseline | at 12 months stimulation
  MADRS: see above
HDRS total score during long-term follow-up compared to baseline | at 12 months stimulation
  see above
CGI total score | at 6 and 12 months DB stimulation compared to baseline
  see above
GAF total score | at 6 and 12 months DB stimulation compared to baseline
  see above
BDI-II total score | at 6 and 12 months DB stimulation compared to baseline
  see above
SF-36 total score | at 6 and 12 months DB stimulation compared to baseline
  see above
Neuropsychological Assessments: Rey Complex Figure Test (CFT) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: d2 concentration test (d2) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: 5-Point-Test | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Wechsler Adult Intelligence Scale (WAIS) (vocabulary, similarities) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Mini-Mental-Status-Test (MMST) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Multiple-Choice Vocabulary Intelligence Test (MWT-B) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Rey Visual Design Learning Test (RVDLT) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Word Fluency Test | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Stroop-Test | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Test for Attentional Performance (TAP) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Trail-Making Test (TMT) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Verbal Memory and Learning Ability Test | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Hopper Visual Organization Test (VOT) | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Neuropsychological Assessments: Digit-Span and Block-Span Test | at 6 months DBS compared to baseline and at end of the study compared to baseline, assessed up to 77 weeks
  see above
Incidence of relapse into clinical depression after tapering down of DBS | From discontinuation of DBS until the date of first documented relapse, assessed up to 12 weeks
  The incidence of relapse into clinical depression after discontinuation of DBS will be assessed.
Pattern of metabolic activity as measured by FDG-PET at 1 week and 4 months after implantation compared to baseline | at 1 week and 4 months after implantation compared to baseline
  Change of metabolic activity in the prefrontal and orbitofrontal cortex as well as in subcortical regions (nucl. accumbens, amygdala) (exploratory endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Schlaepfer, Prof. Dr., Principal Investigator — University Hospital Freiburg
Locations (2):
- Université Grenoble Alpes, Grenoble, France
- University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany